CLINICAL TRIAL: NCT00769730
Title: Evaluation the Possible Influence of Transcatheter Arterial Chemoembolization on Hepatitis B Viral Replication
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Zu-Yau Lin/Kaohsiung Medical University Hospital, Kaohsiung Medical University Hospital
Other Study IDs: KMUH-IRB-960331
Record Dates: First submitted 2008-09-29; First posted 2008-10-09 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-07

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B Virus
Keywords: hepatocellular carcinoma; hepatitis B virus; transcatheter arterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with hepatocellular carcinoma caused by hepatitis B virus who will be treated by transcatheter arterial chemoembolization were included.

SUMMARY:
Transcatheter arterial chemoembolization (TACE) is the traditional method for the palliative management of patients with hepatocellular carcinoma (HCC). Few previous studies had demonstrated that the serum level of anticancer drug from patients treated by TACE was similar to those treated by systemic chemotherapy. Since systemic chemotherapy may have the possibility to influence patient's general defense ability, hepatitis B virus may reactivate after chemotherapy.This study is to investigate the possibility of TACE in the reactivation of hepatitis B virus.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common malignant tumor of the liver. Chronic hepatitis B infection is the common etiology for the development of HCC. Transcatheter arterial chemoembolization (TACE) is the traditional method for the palliative management of patients with HCC. Few previous studies had demonstrated that the serum level of anticancer drug from patients treated by TACE was similar to those treated by systemic chemotherapy. Since systemic chemotherapy may have the possibility to influence patient's general defense ability, hepatitis B virus may reactivate after chemotherapy. There is no study to investigate the possibility of TACE in the reactivation of hepatitis B virus. This project will collect 20 patients with HCC caused by hepatitis B who are planned to be treated by TACE. Quantitative determination of viral load in blood will be performed before TACE, the first and the third month after TACE to investigate the influence of TACE on hepatitis B virus replication. This study will not influence the doctor's decision in the management of HCC and the procedure of TACE. The serum used for HBV DNA examination is concomitantly obtained during regular blood sampling for TACE preparation and follow-up of patient. The amount of blood needed for each time HBV DNA examination is less than 10 ml.

ELIGIBILITY:
Inclusion Criteria:

* patients with hepatocellular carcinoma caused by hepatitis B virus without antiviral drug treatment and patients will be treated by transcatheter arterial chemoembolization

Exclusion Criteria:

* patients already received antiviral drug management

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hepatocellular carcinoma caused by hepatitis B virus who will be treated by transcatheter arterial chemoembolization
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
HBV viral load | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: zu y lin, MD, Ms, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan